CLINICAL TRIAL: NCT00189800
Title: A Study of Solifenacin Succinate Compared to Tolterodine in Patients With Overactive Bladder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 90502/KOoTD01
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2006-10

CONDITIONS: Overactive Bladder
Keywords: Solifenacin; tolterodine; randomized controlled trial; double-blind method
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

INTERVENTIONS:
Drug: Solifenacin succinate

SUMMARY:
The purpose of this study is to ascertain the clinical results of solifenacin succinate of PIII study conducted in the original country using Korean patients with an overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of overactive bladder
* Must be able to complete the micturition diary

Exclusion Criteria:

* Pregnant or lactating
* Clinically significant outflow obstruction
* Significant post void residual urine
* Significant stress incontinence
* Urinary tract infection
* Chronic inflammation
* Bladder stones
* Previous pelvic radiation therapy
* Previous or current malignant disease of the pelvic organs
* Uncontrolled narrow angle glaucoma
* Urinary or gastric retention
* Electrostimulation therapy
* Bladder training
* Diabetic neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Jeong Gu Lee, Principal Investigator — Department of Urology, Korea University Anam Hospital
Locations (10):
- South Korea (10):
  - Anyang
  - Bucheon-si
  - Busan
  - Cheonan
  - Daegu
  - Daejeon
  - Gwangju
  - Incheon
  - Seoul
  - Suwon

REFERENCES:
- [Background] EU Shi-liang, et al. Efficacy and safety of solifenacin in the treatment of patients with urgency and urge incontinence. Chin J Urol (2009) 30(9); 1-5
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Choo MS, Lee JZ, Lee JB, Kim YH, Jung HC, Lee KS, Kim JC, Seo JT, Paick JS, Kim HJ, Na YG, Lee JG. Efficacy and safety of solifenacin succinate in Korean patients with overactive bladder: a randomised, prospective, double-blind, multicentre study. Int J Clin Pract. 2008 Nov;62(11):1675-83. doi: 10.1111/j.1742-1241.2008.01898.x. PMID 19143854